CLINICAL TRIAL: NCT04531748
Title: Selective Estrogen Modulation and Melatonin in Early COVID-19
Acronym: SENTINEL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding
Sponsor: Reena Mehra, MD (Other)
Responsible Party: Sponsor-Investigator, Reena Mehra, MD, Director, Sleep Disorders Research, Neurological Institute, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-842
Record Dates: First submitted 2020-08-27; First posted 2020-08-28 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Covid19
Keywords: covid19; coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Toremifene; Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Medical Safety Officer will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Toremifene + Melatonin (Active Comparator): 100mg oral Melatonin on Days 1 & 2 (40mg in the morning and 60mg in the evening), 60 mg on Days 3-14, (20mg in the morning and 40mg in the evening).
  60mg oral toremifene daily days 1-14.
  Interventions: Drug: Toremifene; Drug: Melatonin
- Melatonin + Placebo (Active Comparator): 100mg oral Melatonin on Days 1 & 2 (40mg in the morning and 60mg in the evening) and 60 mg on Days 3-14, (20mg in the morning and 40mg in the evening).
  Interventions: Drug: Melatonin; Other: Placebo
- Placebo (Placebo Comparator): Oral placebo will be used with the same number and appearance to the pills as the interventions
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Toremifene — Participants will be instructed to take 60mg of oral toremifene capsule daily, 30 minutes before bedtime.
  Arms: Toremifene + Melatonin
Drug: Melatonin — Participants will be instructed to take the pills orally around the same time in the morning and 30 minutes prior to bedtime in the evening.
  Arms: Melatonin + Placebo; Toremifene + Melatonin
Other: Placebo — Oral placebo will be used with the same number and appearance to the pills as the interventions.
  Arms: Melatonin + Placebo; Placebo

SUMMARY:
This study is a randomized, double-blind, controlled clinical trial to evaluate the effects of toremifene and/or melatonin in adults with mild COVID-19.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, controlled clinical trial to evaluate the effects of a 14 day intervention of toremifene plus melatonin or melatonin in adults with mild COVID-19.

The study will evaluate the progression of clinical signs and symptoms (fever, dyspnea, cough, fatigue daily score) and any adverse outcomes in comparison to placebo for 30 days.

The successful completion of this project offers high potential to identify effective treatment (e.g., toremifene plus melatonin and/or melatonin) rapidly for patients with early COVID-19 and to provide, important, fundamental mechanistic insights.

ELIGIBILITY:
Inclusion Criteria:

* Clinical testing positive for SARS-Cov-2 by standard RT-PCR or equivalent test
* Willing and able to give informed consent for participation in the study and agrees with the study and its conduct
* Age>18 years
* Fluency in English or Spanish language, functional literacy
* Able to swallow pills
* COVID-19 Daily Sign and Symptom score of 2-8

Exclusion Criteria:

* History of deep venous thrombosis or pulmonary embolism
* Hypercoagulable disorders (e.g. lupus anticoagulant, deficiency of protein C or S)
* Embolic stroke
* Liver disease
* History of endometrial cancer
* Menopausal hormone therapy or oral, injectable or transdermal contraceptives
* Depression which is not optimally treated (assessed via medical record and patient will be asked if she/he feels that depression is optimally treated)
* Medications which prolong the QT interval (e.g. hydroxychloroquine or azithromycin) or those with long QT syndrome (heritable or acquired). Examples of other medications which prolong the QT interval include: Agents generally accepted to prolong QT interval include Class 1A (e.g., quinidine, procainamide, disopyramide) and Class III (e.g., amiodarone, sotalol, ibutilide, dofetilide) antiarrhythmics; certain antipsychotics (e.g., thioridazine, haloperidol); certain antidepressants (e.g., venlafaxine, amitriptyline); certain antibiotics (e.g., erythromycin, clarithromycin, levofloxacin, ofloxacin); and certain anti-emetics (e.g., ondansetron, granisetron) (Please refer to Appendix for detailed list of medications)
* Inability to participate in follow up assessment
* Dementia/cognitive dysfunction
* Pregnancy (pregnancy testing will be performed to determine eligibility)
* Breastfeeding
* Participating in other COVID-19 trials
* Immunodeficiency (including HIV, Hepatitis C, bone marrow transplant history, on immunosuppressant medications)
* Current hospitalization
* Seizure disorder
* History of rheumatoid arthritis
* Heart failure (NYHA Class III or IV)
* Current diagnosis of renal insufficiency/failure
* QTc >470ms per 12-lead ECG
* Calcium >10.2mg/dL
* AST or ALT > 2x upper limit of normal (ULN)
* D-dimer >= 1000 u/L
* Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2
* On other treatment(s) for COVID-19 (e.g. hydroxychloroquine, remdesivir)
* Anticoagulant medications (e.g. coumadin, glycoprotein IIa/IIIb inhibitors)
* Clinical signs of severe or critical severity of COVID-19 (e.g. shortness of breath at rest, Respiratory rate ≥ 30 per minute, heart rate ≥ 125 per minute, SpO2 ≤ 93% on room air)
* Use of supplemental oxygen
* Moderate to severe pulmonary disease up to PI discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Peak increase in COVID-19 Sign and Symptom score | Screening to 28 days
  Score total of 0-12 assessed daily. Each category based on severity of symptoms of Cough, Shortness of breath, Fatigue/tiredness and daily temperature on a rating scale of 0-3.

SECONDARY OUTCOMES:
Nadir Oxygen Saturation | Day 1 through day 14
  Daily mean values
Peak Heart Rate | Day 1 through day 14
  Daily mean values
Time to COVID-19 Sign and Symptom score resolution | Screening to 28 days
  Score total of 0-12 assessed daily. Each category based on severity of symptoms of Cough, Shortness of breath, Fatigue/tiredness and daily temperature on a rating scale of 0-3.
Time to WHO 7-point ordinal scale score of 3 or higher | Day 1 to Day 30
  1. not hospitalized, no limitation of activities (or resumption of normal activity)
  2. not hospitalized but limitation on activities
  3. hospitalized, not requiring supplemental oxygen
  4. hospitalized, requiring supplemental oxygen (low-flow, e.g., nasal prong)
  5. hospitalized, requiring non-invasive ventilation and/or high-flow oxygen
  6. hospitalized, on invasive ventilation or ECMO
  7. death

CONTACTS AND LOCATIONS:
Overall Officials: Reena Mehra, MD, Principal Investigator — The Cleveland Clinic